CLINICAL TRIAL: NCT03411590
Title: The Effect of Fortified Growing-up Milk on Growth and Micronutrient Status of Nigerian Toddlers
Acronym: GaGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: FrieslandCampina WAMCO Nigeria PLC (Industry)
Collaborators: Lagos State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-GAGA-GND
Record Dates: First submitted 2017-12-11; First posted 2018-01-26 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Malnutrition; Mild; Iron-deficiency Anemia; Nutritional Stunting; Nutritional Wasting; Nutritional Deficiency; Enterobacteriaceae Infections
MeSH Terms: conditions — Malnutrition; Lymphoma, Follicular; Anemia, Iron-Deficiency; Enterobacteriaceae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 200ml (Other): Toddlers will be allocated to the 200 ml group
  Interventions: Other: Fortified milk Powder
- 400ml (Other): Toddlers will be allocated to the 400 ml group
  Interventions: Other: Fortified milk Powder
- 600ml (Other): Toddlers will be allocated to the 600 ml
  Interventions: Other: Fortified milk Powder

INTERVENTIONS:
Other: Fortified milk Powder — Toddlers will be allocated to the 200 ml group and will receive on a daily basis 32g of growing up milk powder respectively, in doses of 16 g, which can be reconstituted with 180 ml water to a final volume of about 200 ml of milk. The intervention period will last for 6 months. For the 200 ml test group, this translates into 32 g of growing up milk powder supply as one dose per day (in the morning)

SUMMARY:
It is well known than an important part of Nigerian children from the lower social economic class have nutrient deficiencies. Fortified products, such as growing up milks (GUM), may play an important role in reducing the risk and incidence of nutrient deficiencies. However, affordability of GUM is an issue.

In this project the effects are studied of different daily intakes of GUM on iron status, growth, several other nutrient status parameters in blood and urine, cognitive development, and the intestinal microbiome in Nigerian toddlers 1-3 years of age.

The project is a collaboration with the department of Paediatrics and Child health of the Lagos State University College of Medicine in Lagos. The design is based on a three-arm, open (partly blind: statistics, biochemical analyses), randomized intervention trial. Recruitment will take place in Ijora-Badia community in Apapa-Iganmu Local Council Development Area (LCDA) in Lagos. The three groups will be given a multi-micronutrient fortified growing-up milk (PEAK), in amounts of 200, 400 or 600 ml per day during a period of 6 months. Primary objective of this study is to reduce iron deficiency anemia. Based on this objective, in total 150 children have to be included in this study.

DETAILED DESCRIPTION:
The present study will be a three-arm, open (partly blind) blind, randomized intervention trial in Nigerian children (12-36 months of age). Recruitment will take place in Ijora-Badia community in Apapa-Iganmu Local Council Development Area (LCDA), Lagos, South-West Nigeria. Ijora-Badia community has the highest burden of under-nutrition; In addition, it consists predominantly of low to middle socioeconomic status population, which is nationally representative, thus making it an ideal choice for this study. All families that are permanent residents of Ijora-Badia and have children aged 12-36 months will be invited to participate in the study. Before screening and recruitment will take place, parents or legal guardians of all potential candidates (toddlers) will be fully informed about the study, requirements and procedures. This means that at the day of screening, recruitment and enrolment, 10-20 children per day, fulfilling inclusion criteria, will be directly assigned to one of the three study groups when a written informed consent is obtained from the parents or legal guardians.

At the day of screening and recruitment, mothers will be required to bring their child to the clinic. At this initial screening toddlers will be evaluated to assess their eligibility for participation to the study according to the inclusion and exclusion criteria (i.e. anthropometric measurements, blood collection for the assessment of haemoglobin levels and information collected by parents). Those toddlers meeting all inclusion criteria will be considered as eligible and will be randomised to one of the three study groups. Prior to the initiation of the intervention, all eligible study participants will be dewormed (medicine, brand, dosage). Baseline measurements will take place that same day, and after 6 months of intervention: anthropometric measurement, a cognitive test (30 minutes), and venous blood sampling (8 ml). For food and nutrient intake indices, and faecal sampling, a proper planning will be made, to be sure that it takes place within 3 days following baseline measurements.

The three groups will be given a multi-micronutrient fortified growing-up milk, in amounts of 200, 400 or 600 ml per day. In case of 400 and 600 ml, the portions (200 ml each) will be spread during the day. Airtight packed portions of milk powder sachets will be delivered weekly at the families by field monitors who also provide instructions for use as well as collect empty sachets for a compliance check. Consumption of test product will start as soon as all baseline examinations and samples have been completed and collected, and will last for 6 months.

Prior to the initiation of the screening and recruitment phase, the study protocol will have to be approved by the Lagos State University Teaching Hospital Research/Ethics Committee, and has to be registered in an acknowledged trial register.

ELIGIBILITY:
Inclusion Criteria:

1. Normal term birth (caesarean section excluded)
2. Boys and girls in the age range of 12 to 36 months at enrolment
3. Apparently healthy at screening (assessed with the use of a medical history record)
4. Hb ≥70 g/L and ≤109 g/L, according to WHO guidelines 27
5. Mild to moderate acute malnutrition (i.e. HAZ, WAZ <-1 SD and > -3 SD)
6. Parents and/or legal guardians are residents of Oshodi LGA
7. Parents and/or legal guardians do not plan to migrate during the study
8. Written informed consent from parents and/or legal guardians
9. Children able to consume a maximum of 96g (= 600 ml) of product per day

Exclusion Criteria:

1. Severe anaemia (Hb<70 g/L) or normal Hb (Hb≥110 g/L)
2. Severe acute malnutrition (HAZ, WAZ <-3 SD) requiring hospitalization
3. Chronic or severe illness requiring hospitalisation and/or special treatment
4. Recent medical history (past 3 months) of serious infections, injuries and/or surgeries
5. Any known allergies or intolerances to milk or milk ingredients
6. Predominantly breast-fed infants or toddlers
7. Consumption of any other fortified foods or supplements
8. Participation to other micronutrient supplementation programmes
9. Participation to any other nutritional study in the last 6 months
10. Participation to another clinical study or receipt of an investigational drug in the last 30 days
11. Indication that they are likely to move within the period of study intervention
12. Family members of employees of the Sponsor or the study site.
13. Use of any prescription medications prior to and/or during the study period for more than or equal to two weeks.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2018-02-05 (Estimated); Primary Completion 2018-09-08 (Estimated); Study Completion 2019-01-24 (Estimated)

PRIMARY OUTCOMES:
Iron deficiency anaemia | 6 Months
  Prevalence of Iron deficiency anaemia as assessed by haemoglobin concentration

SECONDARY OUTCOMES:
Hematocrit | 6 months
  Hematocrit to substantiate the effect of iron supplementation on Hb
Ferritin | 6 months
  ferritin to substantiate the effect of iron supplementation on Hb concentration
plasma concentrations of specific inflammation markers (i.e. C-Reactive) | 6 months
  plasma concentrations of specific inflammation markers (i.e. C-Reactive)
Weight | 6 months
  Body weight for infants up to 24 months old
Serum concentrations of specific micronutrient status | 6 Months
  Serum concentrations of specific micronutrient status indices, such as vitamins, minerals and trace elements.
Parameters of cognitive development | 6 Months
  Parameters of cognitive development such as Memory tests, attention tests,using screening version of the Bayley III Test for Children
Recumbent length | 6 months
  Length in meters and standing height for toddlers from 24 to 36 months old
Plasma concentrations of specific micronutrient status | 6 months
  Plasma concentrations of specific micronutrient status indices, such as vitamins, minerals and trace elements.
Urine concentrations of specific micronutrient status | 6 Months
  Urine concentrations of specific micronutrient status indices, such as vitamins, minerals and trace elements.

OTHER OUTCOMES:
intestinal microbiome | 6 months
  intestinal microbiome in a subpopulation of infants to explore the effect of 2-7 mg of Fe per day (provided as ferrous-sulfate) on the numbers of and changes in Enterobacteriaceae

CONTACTS AND LOCATIONS:
Overall Officials: Idowu O Senbanjo, MBBS, Principal Investigator — LAGOS STATE UNIVERSITY COLLEGE OF MEDICINE

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Senbanjo IO, Owolabi AJ, Oshikoya KA, Hageman JHJ, Adeniyi Y, Samuel F, Melse-Boonstra A, Schaafsma A. Effect of a Fortified Dairy-Based Drink on Micronutrient Status, Growth, and Cognitive Development of Nigerian Toddlers- A Dose-Response Study. Front Nutr. 2022 Apr 27;9:864856. doi: 10.3389/fnut.2022.864856. eCollection 2022. PMID 35571933